CLINICAL TRIAL: NCT01136148
Title: Evaluation of a Medical and Mental Health Unit Compared With Standard Care for Older People Whose Emergency Admission to an Acute General Hospital is Complicated by Concurrent 'Confusion'.
Brief Title: Trial of a Medical and Mental Health Unit for Older People
Acronym: TEAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); Nottingham University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 10004; RP-PG-0407-10147 (Other Grant/Funding Number: NIHR)
Record Dates: First submitted 2010-06-02; First posted 2010-06-03 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Dementia; Confusion; Cognitive Impairment; Delirium
Keywords: Mental Health; Aged; Hospitals, general; Dementia; Delirium; Dementia and confusion
MeSH Terms: conditions — Dementia; Confusion; Cognitive Dysfunction; Delirium; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A Medical and Mental Health Unit (Experimental): A specialist unit for cognitively impaired older patients admitted as a medical emergency to the acute hospital.
  Interventions: Behavioral: A medical and mental health unit
- Standard care wards (Active Comparator): The standard care provided by the acute hospital for cognitively impaired older patients admitted as a medical emergency.
  Interventions: Behavioral: A medical and mental health unit

INTERVENTIONS:
Behavioral: A medical and mental health unit — A specialist medical and mental health unit with both physician and psychiatric medical and nursing staff, and mental health experienced therapists. Emphasis will be on early and accurate diagnosis, multidisciplinary management, rigorous communication and goal setting, discharge planning and interface with community services.

SUMMARY:
This research is an evaluation of the MMHU compared to standard care. Patients who are over 65 and 'confused' at admission will be randomly allocated to the MMHU or standard care. The MMHU does not have capacity for all confused older patients admitted to NUH, and random allocation is similar to what happens in practice currently. For this study, 480 of these patients will be recruited, together with a carer (240 from the MMHU, 240 from standard care wards). The investigators will collect baseline information about the patient participant's physical and mental health and disability.

The investigators will count the total days spent at home and measure patient participants' health status after 3 months, and use of resources over six months. Carer strain and quality of life will be measured at baseline and follow up.

DETAILED DESCRIPTION:
The objectives of this study are:

1. To evaluate whether a specialist multidisciplinary MMHU for older people with 'confusion', admitted to a general hospital as an emergency, is associated with better outcomes than standard care.
2. To study the quality of care on the MMHU compared with standard care
3. To perform a health economic analysis, from the perspective of health and social care.

The principal hypotheses being tested are:

* That care on the MMHU is associated with more days spent at home (in the 3 months after recruitment) than care on standard wards
* That care on the MMHU is associated with better health status measured at 3 months, in terms of quality of life, behavioural disturbance, cognitive function, disability, participation, mortality and care home residence.
* That care on the MMHU is associated with better psychological well being amongst carers and reduced carer strain compared with standard care.
* That the quality of care and patient experience for patients on the MMHU is superior to that on standard care wards.
* That care on the MMHU is cost-effective compared with that on standard care wards.

The setting for the study is a large NHS acute teaching hospital organisation with 2 campuses (Queens Medical Centre and City Hospital), comprising 1800 beds, serving a population of 700 000 for general hospital services.

Sample size is determined by available resources. 240 patients randomised to the MMHU unit over 24 months, and an equal number of controls, should be sufficient to measure, with 80% power, a 3 to 6-day reduction in length of stay, and 15% increase in the proportion of participants discharged home (e.g. 50% to 65%). Power will be greater for scaled outcomes, and the 'days at home' outcome.

The main study will run for up to 24 months from July 2010. Follow up will be 3 months after randomisation.

Prior to trial commencement we will run 1 or 2 short pilot studies, during which we will test the recruitment and ward allocation processes.

The study is designed to be robust, despite being constrained by the operational needs of the clinical service, and both service and research capacity.

The NHS Trust clinical service has agreed that, for the duration of the study, allocation to the MMHU will be by randomisation. This is not part of the research, but represents clinical service support for it. Potential participants will be identified by the Acute Medical Unit, on simple criteria (''confused', over 65'). The MMHU will confirm clinical eligibility and complete a screening log. If there is a bed available on MMHU the patient will be randomised using an internet based randomisation system (with stratification on care home residence), and the patient assigned to MMHU or a standard care ward. Non-randomised patients can be referred, and, if appropriate, randomised, later in their hospital stay.

Research eligible patients and carers will be invited to participate in research, once on their allocated ward. Consent and participation will be for data collection, observation of care, and follow up only. Excluded patients will continue on their allocated ward outside the trial.

ELIGIBILITY:
Inclusion Criteria:

* Patient participants will be over 65, admitted as an emergency to Nottingham University Hospital NHS Trust, with an established or possible physical health problem and concurrent 'confusion', clinically eligible for management on the Medical and Mental Health Unit.
* Carer participants will be a family member or carer, in regular contact with the patient participant, to serve both as an informant, and, and to study carer health and outcomes.
* Confusion will be loosely defined, including working diagnoses of:
* Delirium
* Dementia
* Dementia with a suspicion of super-added delirium

Exclusion Criteria:

* Those who require sectioning under the Mental Health Act
* Those with intoxication to illicit drugs or alcohol, or the immediate care of patients with overdose
* Those with a primary psychiatric problem in the absence of suspected significant physical or functional co-morbidity.
* Those who are severely medically ill, requiring intensive monitoring or therapy (critical care), or sub-specialist medical intervention (e.g. severe acute GI bleeding, respiratory support).
* Those with an overriding clinical need for management in another service e.g. stroke, orthogeriatric, renal, oncology.
* Those with personality disorder, depression or anxiety as the primary psychiatric diagnosis.
* Those who are registered with a non - Nottingham Primary Care Trust General Practitioner.
* Those who do not speak English and have no family translator.

Ages: 65 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 600 (Actual)
Dates: Start 2010-07; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Number of days at home in the 3 months after randomisation | 3 months
  The primary outcome will be number of days spent at home in the three months following recruitment (or remaining in a care home for those previously resident at recruitment). This encompasses mortality, discharge, length of hospital stay, and ability to sustain discharge and avoid readmission. 'Days at home' will be calculated as 90 days minus the nuimber of days spent dead, in residential intermediate care units, in hospital, in respite care or in a new care home placement at a higher level of dependency.

SECONDARY OUTCOMES:
Quality of life | 3 months
  Dementia quality of life (Demqol, patient and proxy) and generic quality of life (Euroqol EQ5D).
Behavioural disability | 3 months
  Neuropsychiatric inventory.
Mortality | 3 month
Personal activities of daily living | 3 months
  Barthel ADL Index
Participant / generic disability | 3 months
  short London Handicap Scale
Cognition | 3 months
  MMSE, in particular to detect recovery of delirium
Carer satisfaction with hospital care | 1-3 weeks post discharge from index admission
  Satisfaction with care received questionnaire
Carer strain and general health | 3 months
  Carer strain index and carer general health questionnaire GHQ-12.
Service Outcomes | 3 months
  Days in each type of ward. Hospital re-admissions, and total hospital length of stay. New institutionalisation (or moving to a higher level of dependency for those in a care home) Days in a care home (including respite care) GP visits, and use of other primary care contacts (district nurse, community matron, practice nurse) Hospital appointments Attendances at physical and mental health day hospitals Contact with community mental health teams (including community psychiatric nursing) Use of ambulance service Use of social service home care and day centres.
Quality of care and patient experience on the ward | During hospital stay.
  Quality of care and patient experience will be measured using Dementia Care Mapping on both the MMHU and standard care. Dementia Care Mapping provides a structured record of activity levels, mood and engagement of participants and the quality of staff interactions over a 4-6 hour period.
Health and social care costs | 3 months
  Service outcomes will be costed using specific costs where available or standard reference costs otherwise.

CONTACTS AND LOCATIONS:
Overall Officials: John R Gladman, Principal Investigator — University of Nottingham
Locations (1):
- Nottingham University Hospitals NHS Trust, Nottingham, Nottingham, United Kingdom

REFERENCES:
- [Derived] Tanajewski L, Franklin M, Gkountouras G, Berdunov V, Harwood RH, Goldberg SE, Bradshaw LE, Gladman JR, Elliott RA. Economic Evaluation of a General Hospital Unit for Older People with Delirium and Dementia (TEAM Randomised Controlled Trial). PLoS One. 2015 Dec 18;10(12):e0140662. doi: 10.1371/journal.pone.0140662. eCollection 2015. PMID 26684872
- [Derived] Goldberg SE, Whittamore KH, Pollock K, Harwood RH, Gladman JR. Caring for cognitively impaired older patients in the general hospital: a qualitative analysis of similarities and differences between a specialist Medical and Mental Health Unit and standard care wards. Int J Nurs Stud. 2014 Oct;51(10):1332-43. doi: 10.1016/j.ijnurstu.2014.02.002. Epub 2014 Feb 15. PMID 24613652
- [Derived] Goldberg SE, Bradshaw LE, Kearney FC, Russell C, Whittamore KH, Foster PE, Mamza J, Gladman JR, Jones RG, Lewis SA, Porock D, Harwood RH; Medical Crises in Older People Study Group. Care in specialist medical and mental health unit compared with standard care for older people with cognitive impairment admitted to general hospital: randomised controlled trial (NIHR TEAM trial). BMJ. 2013 Jul 2;347:f4132. doi: 10.1136/bmj.f4132. PMID 23819964
- [Derived] Harwood RH, Goldberg SE, Whittamore KH, Russell C, Gladman JR, Jones RG, Porock D, Lewis SA, Bradshaw LE, Elliot RA; Medical Crises in Older People Study Group (MCOP). Evaluation of a Medical and Mental Health Unit compared with standard care for older people whose emergency admission to an acute general hospital is complicated by concurrent 'confusion': a controlled clinical trial. Acronym: TEAM: Trial of an Elderly Acute care Medical and mental health unit. Trials. 2011 May 13;12:123. doi: 10.1186/1745-6215-12-123. PMID 21569471